CLINICAL TRIAL: NCT02963376
Title: A Phase Ib/II Dose-finding Study of DDFPe in Patients With Acute Ischemic Stroke
Brief Title: A Phase Ib/II in Patients With Acute Ischemic Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NuvOx LLC (Industry)
Collaborators: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 205529
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Results first posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-08

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 0.05 mL/kg DDFPe (Active Comparator): This study is a randomized, placebo controlled, blinded escalating dose study designed to determine the maximum tolerated dose to intravenous administration of DDFPe. At each of the three dose levels 0.10, 0.17 mL/kg) six subjects will receive DDFPe and two will receive placebo.
  Interventions: Drug: 0.05 mL/kg DDFPe
- 0.05 mL/kg Placebo (Placebo Comparator): This study is a randomized, placebo controlled, blinded escalating dose study designed to determine the maximum tolerated dose to intravenous administration of DDFPe. At each of the three dose levels 0.10, 0.17 mL/kg) six subjects will receive DDFPe and two will receive placebo.
  Interventions: Drug: 0.05 mL/kg Placebo
- 0.10 mL/kg DDFPe (Active Comparator): This study is a randomized, placebo controlled, blinded escalating dose study designed to determine the maximum tolerated dose to intravenous administration of DDFPe. At each of the three dose levels 0.10, 0.17 mL/kg) six subjects will receive DDFPe and two will receive placebo.
  Interventions: Drug: 0.10 mL/kg DDFPe
- 0.10 mL/kg Placebo (Placebo Comparator): This study is a randomized, placebo controlled, blinded escalating dose study designed to determine the maximum tolerated dose to intravenous administration of DDFPe. At each of the three dose levels 0.10, 0.17 mL/kg) six subjects will receive DDFPe and two will receive placebo.
  Interventions: Drug: 0.10 mL/kg Placebo
- 0.17 mL/kg DDFPe (Active Comparator): This study is a randomized, placebo controlled, blinded escalating dose study designed to determine the maximum tolerated dose to intravenous administration of DDFPe. At each of the three dose levels 0.10, 0.17 mL/kg) six subjects will receive DDFPe and two will receive placebo.
  Interventions: Drug: 0.17 mL/kg DDFPe
- 0.17 mL/kg Placebo (Placebo Comparator): This study is a randomized, placebo controlled, blinded escalating dose study designed to determine the maximum tolerated dose to intravenous administration of DDFPe. At each of the three dose levels 0.10, 0.17 mL/kg) six subjects will receive DDFPe and two will receive placebo.
  Interventions: Drug: 0.17 mL/kg Placebo

INTERVENTIONS:
Drug: 0.05 mL/kg DDFPe — Prior to injection, DDFPe will be prepared by pharmacy staff. DDFPe will be administered based on weight. Each dose will be prepared on the day of administration and infused directly into the patient using a slow i.v push. The i.v. push shall be 5-10 minutes in duration. DDFPe dosage volume in cc for 0.05 mL/kg based on patient body weight in kilograms (kg).
  Other Names: Dodecafluoropentane emulsion (DDFPe), NanO2TM
  Arms: 0.05 mL/kg DDFPe
Drug: 0.05 mL/kg Placebo — Prior to injection, the placebo will be prepared by pharmacy staff. The placebo will be administered based on weight at designated doses Each dose will be prepared on the day of administration and infused directly into the patient using a slow i.v push. The i.v. push shall be 5-10 minutes in duration. The placebo dosage volume in cc for 0.05 mL/kg is based on patient body weight in kilograms (kg).
  Arms: 0.05 mL/kg Placebo
Drug: 0.10 mL/kg DDFPe — Prior to injection, DDFPe will be prepared by pharmacy staff. DDFPe will be administered based on weight at designated doses. Each dose will be prepared on the day of administration and infused directly into the patient using a slow i.v push. The i.v. push shall be 5-10 minutes in duration. DDFPe dosage volume in cc for 0.10 mL/kg based on patient body weight in kilograms (kg).
  Other Names: Dodecafluoropentane emulsion (DDFPe), NanO2TM
  Arms: 0.10 mL/kg DDFPe
Drug: 0.10 mL/kg Placebo — Prior to injection, the placebo will be prepared by pharmacy staff. The placebo will be administered based on weight at designated doses. Each dose will be prepared on the day of administration and infused directly into the patient using a slow i.v push. The i.v. push shall be 5-10 minutes in duration. The placebo dosage volume in cc for 0.10 mL/kg is based on patient body weight in kilograms (kg).
  Arms: 0.10 mL/kg Placebo
Drug: 0.17 mL/kg DDFPe — Prior to injection, DDFPe will be prepared by pharmacy staff. DDFPe will be administered based on weight at designated doses. Each dose will be prepared on the day of administration and infused directly into the patient using a slow i.v push. The i.v. push shall be 5-10 minutes in duration. DDFPe dosage volume in cc for 0.17 mL/kg based on patient body weight in kilograms (kg).
  Other Names: Dodecafluoropentane emulsion (DDFPe), NanO2TM
  Arms: 0.17 mL/kg DDFPe
Drug: 0.17 mL/kg Placebo — Prior to injection, the placebo will be prepared by pharmacy staff. The placebo will be administered based on weight at designated doses. Each dose will be prepared on the day of administration and infused directly into the patient using a slow i.v push. The i.v. push shall be 5-10 minutes in duration. The placebo dosage volume in cc for 0.17 mL/kg is based on patient body weight in kilograms (kg).
  Arms: 0.17 mL/kg Placebo

SUMMARY:
Stroke is the fifth leading cause of death in the United States and is the leading cause of long term disability. Distinct geographic disparities in stroke mortality, with highest rates in the southeast United States including Arkansas, are known as the "stroke belt." There the average stroke mortality is ≈20% to 40% higher than the rest of the nation. Stroke is the leading cause of serious long-term disability. Between 2012 and 2030, disability and medical costs related to stroke are projected to triple, from $71.6 billion to $184.1 billion, with the majority of the projected increase in costs arising from those 65 to 79 years of age.

There are two main forms of stroke, ischemic and hemorrhagic. An ischemic stroke occurs in 85% of cases and is caused by cerebral vessel occlusion, obstructing blood flow to a portion of the brain. Currently, the only approved therapies for acute ischemic stroke are IV tissue plasminogen activator (tPA), a thrombolytic agent that clears the thrombus within the blood vessel, or intra-arterial catheter thrombectomy. Despite the availability of therapy, it reaches only approximately 7% of ischemic stroke victims in the United States5. Delay beyond the effective time window for therapy is a common reason for failure.

To reduce the devastating impact of stroke on individuals and society, the investigators continue to seek ways to improve functional recovery and limit ischemic damage in stroke patients. The potential neuroprotective agent, dodecafluoropentane emulsion (DDFPe) has recently shown strong positive effects in pre-clinical animal models of acute ischemic stroke6-11. Other perfluorocarbons have been tested in humans as potential neuroprotectants and blood substitutes yet none have been successful.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-80 years
* Diagnosis of AIS
* Body weight ≥ 45 kg
* NIHSS between 2 and 20
* Patient or legal authorized representative (LAR) must be willing and able to understand the study and provide written informed consent

Exclusion Criteria:

Currently pregnant or breastfeeding

* History of significantly impaired renal or hepatic function
* Hemorrhage or hemorrhagic stroke on CT scan
* Prior stroke, intracranial surgery, or major head trauma within three months prior to enrollment
* Pre-stroke modified Rankin Scale (mRS) ≥ 2
* Myocardial infarction within six (6) months prior to enrollment
* Unstable angina, New York Heart Association (NYHA) Class II or greater congestive heart failure
* Uncontrolled hypertension (SBP > 180 and/or diastolic blood pressure (DBP) > 110 mmHg)
* Known long QT syndrome or QTc > 450 milliseconds (ms) in males and > 470 ms in females
* Uncontrolled arrhythmia or history of clinically significant arrhythmia within the past six (6) months (except atrial fibrillation)
* Clinically significant chronic obstructive pulmonary disease (COPD) or other pulmonary condition that is not controlled by medication or requires oxygen frequently or continuously
* Pneumonia, bronchitis, or other acute respiratory disease
* Current anticoagulant therapy except for antiplatelet therapy (aspirin, NSAIDs) and prophylactic doses of low molecular weight heparin to prevent deep vein thrombosis. Note: tPA administered as part of subjects' therapy for AIS is allowed.
* History of allergic reaction attributed to compounds of similar chemical composition to DDFPe (see Investigator's Brochure).
* Subject has received any investigational drug within thirty (30) days prior to enrollment into the study
* Inability to comply with the study procedures
* History or evidence of any other clinically significant condition that, in the opinion of the investigator, might pose a safety risk to subjects or interfere with study procedures, evaluation, or completion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2018-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Culp, MD, Principal Investigator — University of Arkansas; Sanjeeva Onteddu, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Result] Culp WC, Onteddu SS, Brown A, Nalleballe K, Sharma R, Skinner RD, Witt T, Roberson PK, Marsh JD. Dodecafluoropentane Emulsion in Acute Ischemic Stroke: A Phase Ib/II Randomized and Controlled Dose-Escalation Trial. J Vasc Interv Radiol. 2019 Aug;30(8):1244-1250.e1. doi: 10.1016/j.jvir.2019.04.020. PMID 31349978
- See also: Dodecafluoropentane Emulsion in Acute Ischemic Stroke: A Phase Ib/II Randomized and Controlled Dose-Escalation Trial — https://pubmed.ncbi.nlm.nih.gov/31349978/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the study period, 26 patients or their legal authorized representatives were contacted and agreed to participate. Of these, 24 give written informed consent and were included in the study.
Groups:
- 0.05 mL/kg DDFPe: This study is a randomized, placebo controlled, blinded escalating dose study designed to determine the maximum tolerated dose to intravenous administration of DDFPe. At each of the three dose levels (0.05, 0.10, 0.17 mL/kg) six subjects will receive DDFPe and two will receive placebo.
  0.05 mL/kg DDFPe: Prior to injection, DDFPe will be prepared by pharmacy staff. DDFPe will be administered based on weight. Each dose will be prepared on the day of administration and infused directly into the patient using a slow i.v push. The i.v. push shall be 5-10 minutes in duration. DDFPe dosage volume in cc for 0.05 mL/kg based on patient body weight in kilograms (kg).
- 0.05 mL/kg Placebo: This study is a randomized, placebo controlled, blinded escalating dose study designed to determine the maximum tolerated dose to intravenous administration of DDFPe. At each of the three dose levels (0.05, 0.10, 0.17 mL/kg) six subjects will receive DDFPe and two will receive placebo.
  0.05 mL/kg Placebo: Prior to injection, the placebo will be prepared by pharmacy staff. The placebo will be administered based on weight at designated doses Each dose will be prepared on the day of administration and infused directly into the patient using a slow i.v push. The i.v. push shall be 5-10 minutes in duration. The placebo dosage volume in cc for 0.05 mL/kg is based on patient body weight in kilograms (kg).
- 0.10 mL/kg DDFPe: This study is a randomized, placebo controlled, blinded escalating dose study designed to determine the maximum tolerated dose to intravenous administration of DDFPe. At each of the three dose levels (0.05, 0.10, 0.17 mL/kg) six subjects will receive DDFPe and two will receive placebo.
  0.10 mL/kg DDFPe: Prior to injection, DDFPe will be prepared by pharmacy staff. DDFPe will be administered based on weight at designated doses. Each dose will be prepared on the day of administration and infused directly into the patient using a slow i.v push. The i.v. push shall be 5-10 minutes in duration. DDFPe dosage volume in cc for 0.10 mL/kg based on patient body weight in kilograms (kg).
- 0.10 mL/kg Placebo: This study is a randomized, placebo controlled, blinded escalating dose study designed to determine the maximum tolerated dose to intravenous administration of DDFPe. At each of the three dose levels (0.05, 0.10, 0.17 mL/kg) six subjects will receive DDFPe and two will receive placebo.
  0.10 mL/kg Placebo: Prior to injection, the placebo will be prepared by pharmacy staff. The placebo will be administered based on weight at designated doses. Each dose will be prepared on the day of administration and infused directly into the patient using a slow i.v push. The i.v. push shall be 5-10 minutes in duration. The placebo dosage volume in cc for 0.10 mL/kg is based on patient body weight in kilograms (kg).
- 0.17 mL/kg DDFPe: This study is a randomized, placebo controlled, blinded escalating dose study designed to determine the maximum tolerated dose to intravenous administration of DDFPe. At each of the three dose levels (0.05, 0.10, 0.17 mL/kg) six subjects will receive DDFPe and two will receive placebo.
  0.17 mL/kg DDFPe: Prior to injection, DDFPe will be prepared by pharmacy staff. DDFPe will be administered based on weight at designated doses. Each dose will be prepared on the day of administration and infused directly into the patient using a slow i.v push. The i.v. push shall be 5-10 minutes in duration. DDFPe dosage volume in cc for 0.17 mL/kg based on patient body weight in kilograms (kg).
- 0.17 mL/kg Placebo: This study is a randomized, placebo controlled, blinded escalating dose study designed to determine the maximum tolerated dose to intravenous administration of DDFPe. At each of the three dose levels (0.05, 0.10, 0.17 mL/kg) six subjects will receive DDFPe and two will receive placebo.
  0.17 mL/kg Placebo: Prior to injection, the placebo will be prepared by pharmacy staff. The placebo will be administered based on weight at designated doses. Each dose will be prepared on the day of administration and infused directly into the patient using a slow i.v push. The i.v. push shall be 5-10 minutes in duration. The placebo dosage volume in cc for 0.17 mL/kg is based on patient body weight in kilograms (kg).
Period: Overall Study
Arm/Group | 0.05 mL/kg DDFPe | 0.05 mL/kg Placebo | 0.10 mL/kg DDFPe | 0.10 mL/kg Placebo | 0.17 mL/kg DDFPe | 0.17 mL/kg Placebo
Started | 6 | 2 | 6 | 2 | 6 | 2
Completed | 6 | 2 | 6 | 2 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: At each of the three dose levels (0.05, 0.10, 0.17 mL/kg) six subjects received DDFPe and two received placebo in this study.
  For this reason, all control subjects are grouped.
Groups:
- Controls (n=6): This study is a randomized, placebo controlled, blinded escalating dose study designed to determine the maximum tolerated dose to intravenous administration of DDFPe. At each of the three dose levels (0.05, 0.10, 0.17 mL/kg) six subjects will receive DDFPe and two will receive placebo.
  For analysis, all control subjects are grouped.
- DDFPe - 0.05 mL/kg (n=6); DDFPe - 0.10 mL/kg (n=6); DDFPe - 0.17 mL/kg (n=6): This study is a randomized, placebo controlled, blinded escalating dose study designed to determine the maximum tolerated dose to intravenous administration of DDFPe. At each of the three dose levels (0.05, 0.10, 0.17 mL/kg) six subjects will receive DDFPe and two will receive placebo.
- Total: Total of all reporting groups
Arm/Group | Controls (n=6) | DDFPe - 0.05 mL/kg (n=6) | DDFPe - 0.10 mL/kg (n=6) | DDFPe - 0.17 mL/kg (n=6) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (7.1) | 61.2 (4.4) | 53.2 (4.8) | 56.2 (4.6) | 56.6 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 2 | 7
  Male | 5 | 4 | 4 | 4 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 1 | 3
  White | 5 | 5 | 6 | 5 | 21
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 6 | 6 | 24
NIHSS Assessment [Median (Full Range); unit: units on a scale] — The NIH Stroke Scale (NIHSS) is an assessment tool that provides a quantitative measure of stroke-related neurologic deficit. The NIHSS is a 15-item neurologic examination. Ratings for each item are scored on a 3- to 5-point scale with 0 as normal. Scores range from 0 to 42, with higher scores indicating greater severity.
  units on a scale | 9.5 [3 to 17] | 6.5 [0 to 12] | 8 [4 to 13] | 4 [2 to 14] | 6.5 [0 to 17]

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of DDFPe Evaluated by Number of Dose Limiting Toxicities
Description: The primary objective of this study is to establish the Maximum Tolerated Dose (MTD) of DDFPe given intravenously at intervals of 90 ± 10 minutes x 3 doses within 12 hours after subjects have had a documented Acute Ischemic Stroke (AIS). The algorithm for determining the MTD is based on the number of subjects who experience a Dose Limiting Toxicity (DLT) in each cohort, as defined in the clinical protocol. If three or more subjects who received DDFPe in an 8 subject cohort experience a DLT, the MTD will be determined to have been exceeded and further enrollment in the cohort as well as dose escalation will stop.
Time Frame: 12 hours after subjects have had a documented Acute Ischemic Stroke (AIS)
Population: No signs of dose-limiting episodes were identified at any dose level, and no MTD was defined.
Measure: Number; unit: Dose Limiting Toxicities
Arm/Group | 0.05 mL/kg DDFPe | 0.05 mL/kg Placebo | 0.10 mL/kg DDFPe | 0.10 mL/kg Placebo | 0.17 mL/kg DDFPe | 0.17 mL/kg Placebo
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2
Dose Limiting Toxicities | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: NIHSS Assessment
Description: The NIH Stroke Scale (NIHSS) is an assessment tool that provides a quantitative measure of stroke-related neurologic deficit. The NIHSS is a 15-item neurologic examination. Ratings for each item are scored on a 3- to 5-point scale with 0 as normal. Scores range from 0 to 42, with higher scores indicating greater severity.
Time Frame: NIHSS scores were recorded at outside hospitals when appropriate and also at the study center as inside baseline NIHSS score. Repeat NIHSS scores were recorded at 2, 3.5, and 7.5 hours after drug injection and on discharge.
Population: At each of the three dose levels (0.05, 0.10, 0.17 mL/kg) six subjects received DDFPe and two received placebo in this study.
  All control subjects are grouped for the NIHSS results. DDFPe results are shown separately for each cohort as well as combined.
Measure: Median (Full Range); unit: units on a scale
Groups:
- Controls (n=6): This study is a randomized, placebo controlled, blinded escalating dose study designed to determine the maximum tolerated dose to intravenous administration of DDFPe. At each of the three dose levels 0.10, 0.17 mL/kg) six subjects will receive DDFPe and two will receive placebo.
  All control patients are grouped for the NIHSS results.
- DDFPe (n=18): This study is a randomized, placebo controlled, blinded escalating dose study designed to determine the maximum tolerated dose to intravenous administration of DDFPe. At each of the three dose levels 0.10, 0.17 mL/kg) six subjects will receive DDFPe and two will receive placebo.
  This column groups the NIHSS results of all DDFPe treated patients.
Arm/Group | Controls (n=6) | DDFPe (n=18) | 0.05 mL/kg DDFPe | 0.10 mL/kg DDFPe | 0.17 mL/kg DDFPe
Number analyzed (Participants) | 6 | 18 | 6 | 6 | 6
units on a scale
  Baseline (PreRx) | 9.5 [3 to 17] | 6.5 [0 to 14] | 6.5 [0 to 12] | 8 [4 to 13] | 4 [2 to 14]
  2 hours | 8 [3 to 17] | 5 [0 to 15] | 6 [0 to 14] | 6.5 [1 to 15] | 2 [0 to 6]
  3.5 hours | 5.5 [3 to 14] | 4.5 [0 to 15] | 5.5 [0 to 12] | 7 [1 to 15] | 2.5 [0 to 5]
  7.5 hours | 4.5 [2 to 14] | 2.5 [0 to 13] | 5.5 [0 to 9] | 5.5 [1 to 13] | 2 [0 to 4]
  Day 7 or Day of Discharge | 3.5 [1 to 11] | 1 [0 to 11] | 2 [0 to 5] | 4 [0 to 11] | 1 [0 to 2]

3. Secondary Outcome: Modified Rankin Scale (mRS)
Description: The modified Rankin Scale is a measure of the degree of disability in patients who have had a stroke with 0 being no symptoms at all to 6 being death. Thus, a higher score indicates greater severity.
Time Frame: mRS values were obtained on Day 7 or Day of Discharge, Day 30 and Day 90.
Population: At each of the three dose levels (0.05, 0.10, 0.17 mL/kg) six subjects received DDFPe and two received placebo in this study.
  All control subjects are grouped for the mRS results. DDFPe results are shown separately for each cohort as well as combined.
Measure: Median (Full Range); unit: units on a scale
Groups:
- Controls (n=6): This study is a randomized, placebo controlled, blinded escalating dose study designed to determine the maximum tolerated dose to intravenous administration of DDFPe. At each of the three dose levels 0.10, 0.17 mL/kg) six subjects will receive DDFPe and two will receive placebo.
  All control patients are grouped for the mRS results.
- DDFPe (n=18): This study is a randomized, placebo controlled, blinded escalating dose study designed to determine the maximum tolerated dose to intravenous administration of DDFPe. At each of the three dose levels 0.10, 0.17 mL/kg) six subjects will receive DDFPe and two will receive placebo.
  This column groups the mRS results of all DDFPe treated patients.
Arm/Group | Controls (n=6) | DDFPe (n=18) | 0.05 mL/kg DDFPe | 0.10 mL/kg DDFPe | 0.17 mL/kg DDFPe
Number analyzed (Participants) | 6 | 18 | 6 | 6 | 6
units on a scale
  Day 7 or Day of Discharge | 2 [1 to 4] | 2 [0 to 4] | 2 [0 to 3] | 3 [0 to 4] | 1.5 [0 to 2]
  30 day | 2.5 [1 to 6] | 1 [0 to 6] | 2 [0 to 6] | 2 [0 to 4] | 0 [0 to 1]
  90 day | 3 [0 to 6] | 1 [0 to 6] | 1.5 [0 to 6] | 2 [0 to 3] | 0 [0 to 1]

ADVERSE EVENTS:
Time Frame: The study treatment follow-up was within 90 days following the last administration of study treatment.
Description: At each of the three dose levels (0.05, 0.10, 0.17 mL/kg) six subjects received DDFPe and two received placebo in this study.
  For this reason, all control subjects are grouped.
Groups:
- Controls (n=6): This study is a randomized, placebo controlled, blinded escalating dose study designed to determine the maximum tolerated dose to intravenous administration of DDFPe. At each of the three dose levels (0.05, 0.10, 0.17 mL/kg) six subjects will receive DDFPe and two will receive placebo.
  For this reason, all control subjects are grouped.
- DDFPe - 0.17 mL/kg; DDFPe Total (n=18): This study is a randomized, placebo controlled, blinded escalating dose study designed to determine the maximum tolerated dose to intravenous administration of DDFPe. At each of the three dose levels (0.05, 0.10, 0.17 mL/kg) six subjects will receive DDFPe and two will receive placebo.
Arm/Group | Controls (n=6) | DDFPe - 0.05 mL/kg (n=6) | DDFPe - 0.10 mL/kg (n=6) | DDFPe - 0.17 mL/kg | DDFPe Total (n=18)
All-Cause Mortality (participants affected / at risk) | 1/6 | 1/6 | 0/6 | 0/6 | 1/18
Serious Adverse Events (participants affected / at risk) | 3/6 | 1/6 | 0/6 | 0/6 | 1/18
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 3/6 | 15/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Controls (n=6) (N=6) | DDFPe - 0.05 mL/kg (n=6) (N=6) | DDFPe - 0.10 mL/kg (n=6) (N=6) | DDFPe - 0.17 mL/kg (N=6) | DDFPe Total (n=18) (N=18)
Confusional State (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac Pacemaker Replacement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular Accident, Secondary Stroke (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Controls (n=6) (N=6) | DDFPe - 0.05 mL/kg (n=6) (N=6) | DDFPe - 0.10 mL/kg (n=6) (N=6) | DDFPe - 0.17 mL/kg (N=6) | DDFPe Total (n=18) (N=18)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arrythmia (Cardiac disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (4)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Electrocardiogram Abnormal (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Infusion Related Reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 2 (4)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vascular device occlusion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Akathisia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (2) | 2 (3) | 0 (0) | 3 (5)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Carotid Endarterectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 2 (5) | 0 (0) | 0 (0) | 2 (5)
Haemorrhoids (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (6) | 2 (2) | 0 (0) | 4 (8)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of the current study primarily concern the exploratory aim toward efficacy, which was greatly underpowered for any purpose other than designing the next study. As with any phase I trial, the small number of cases may only demonstrate side effects and complications that are common.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT02963376/Prot_SAP_000.pdf